CLINICAL TRIAL: NCT05192746
Title: Radial Extracorporeal Shock Wave Therapy Versus High Power Pain Threshold Ultrasound Therapy on Pain,Pressure Threshold Supraspinatus Trigger Point
Brief Title: Radial Extracorporeal Shock Wave Therapy Versus High Power Pain Threshold Ultrasound Therapy in Supraspinatus Tendinitis
Acronym: RESWTHPPTU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hayam Hamza, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/120/03319
Record Dates: First submitted 2021-10-27; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Supraspinatus Tendinitis
Keywords: extracorporeal shock wave; high power pain threshold ultrasound
MeSH Terms: interventions — Control Groups; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: pre post intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A "Control group" (Experimental): Twenty two patients will receive conventional treatment hot pack and exercise (control group).
  .
  Interventions: Other: control group
- group B"Extracorporeal shock wave group": (Experimental): Twenty two patients will receive Radial Extra corporeal Shock Wave Therapy plus conventional treatment hot pack and exercise.
  Interventions: Device: extracorporeal shock wave therapy
- Group C"High power pain threshold ultrasound group": (Experimental): Twenty two patients will receive High-Power Pain Threshold Ultrasound therapy plus conventional treatment hot pack and exercise
  Interventions: Device: high power pain threshold ultrasound

INTERVENTIONS:
Other: control group — Exercise Therapy and hot pack This tendon exercise program is very effective if done consistently. There are five steps to the program: warm up, stretching exercise, strengthening exercise, stretching exercise, and heat.
  Arms: group A "Control group"
Device: extracorporeal shock wave therapy — Shock Master 500 device will be applied once a week for four weeks in total. Each treatment consists of 2000 shocks 3 bar pressure, 20 Hz. Each rESWT session will take about 10 minutes. rESWT application will be performed on the supraspinatus trigger point. In successive treatments, there will be using of an energy density equal to 0.28 mJ/mm2
  Arms: group B"Extracorporeal shock wave group":
Device: high power pain threshold ultrasound — High-power, pain-threshold, ultrasound therapy application (in W/cm2) in continuousmodes, to elicit threshold pain, the ultrasound probe must be kept static on the tendon.
  Intensity will be gradually increased to the level of maximum pain the patient could bear. It will be kept at that level for 4 to 5 seconds and then will be reduced to the half-intensitylevel for another 15 seconds. This procedure will be repeated 3 times.High-power,
  Arms: Group C"High power pain threshold ultrasound group":

SUMMARY:
Extra corporeal shock wave therapy is a treatment method in which high-amplitude sound waves are focused on the targeted body tissue Recently, Extra corporeal shock wave therapy has been proposed as an alternative treatment in patients not responding to pharmaceutical treatment.High power pain threshold ultrasound is the use of therapeutic ultrasound in a continuous mode; with the probe placed directly on affected area (supraspinatus tendon)

DETAILED DESCRIPTION:
Shock wave therapy is an effective method of dissolving calcification and stimulating tissue healing. Extra corporeal shock wave therapy is a treatment method in which high-amplitude sound waves are focused on the targeted body tissue Recently, Extra corporeal shock wave therapy has been proposed as an alternative treatment in patients not responding to pharmaceutical treatment.US have been widely used for more than 40 years in the treatment of musculoskeletal disorders such as tendinitis, tenosynovitis, epicondylitis, bursitis and osteoarthritis. High power pain threshold ultrasound is the use of therapeutic ultrasound in a continuous mode; with the probe placed directly on affected area (supraspinatus tendon) "the intensity of ultrasound is first increased to the threshold pain level (to 1.5 W/cm) and then reduced to one half of that intensity. It was kept at that level for 4 to 5 seconds and then reduced to the half-intensity level for another 15 seconds .

ELIGIBILITY:
Inclusion Criteria:

* Patients' age ranges from 30 to 50 years old.
* Patients are males and females.
* BMI of all subjects were <30 Kg/m2.
* Patients will be diagnosed as supraspinatus tendinitis.
* All patients are medically stable.
* All patients should be conscious and ambulant.
* Patients don't have any nervous system problems
* Patients don't have shoulder disorder other than tendenities
* Patients that didn't undergo any surgery in shoulder joint

Exclusion Criteria:

* • Patients who received intra articular injection from duration less than 3 months.

  * Patients with supraspinatus tendonitis secondary to trauma.
  * Patients with metal implants.
  * Patient who had malignancy in the affected area.
  * Patient with acute infection in the treated area.
  * Diabetic patients
  * Bone infection
  * Shoulder instability
  * Epilepsy
  * Coagulation diseases
  * Rheumatological diseases (rheumatoid arthritis and gouty arthritis)

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 66 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
1. pain intensity[Time Frame:] | up to four weeks
  pain will be measured by visual analogue scale higher score mean worse outcome ten centimeter line from zero to ten, zero mean no pain and ten mean maximum pain
2.range of motion | up to four weeks
  range of motion will be measured by gravititional inclinometer

IPD SHARING:
Plan to Share IPD: No